CLINICAL TRIAL: NCT02023385
Title: Evaluation of the BTL-9000 Low Level Laser Therapy for the Waist Circumferential Reduction
Brief Title: BTL-9000 Low Level Laser Therapy for the Waist Circumferential Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BTL Industries Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BTL-9000 LLLT
Record Dates: First submitted 2013-12-20; First posted 2013-12-30 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2013-12

CONDITIONS: Circumferential Reduction; Waist Circumferential Reduction
Keywords: Low Level Laser Therapy; LLLT; Waist circumferential reduction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LLLT group (Experimental): Subjects in the Low Level Laser Therapy (LLLT) group will be treated with the BTL-9000 LLLT
  Interventions: Device: BTL-9000 LLLT
- Placebo group (Placebo Comparator): Subjects in the Placebo group with be treated with the sham BTL-9000 LLLT
  Interventions: Device: sham BTL-9000 LLLT

INTERVENTIONS:
Device: BTL-9000 LLLT — Irradiation of adipocyte cells within the fat layer with BTL-9000 LLLT for the release of fat and lipids from these cells
  Other Names: BTL-9000 LowLevel Laser Therapy
  Arms: LLLT group
Device: sham BTL-9000 LLLT — Irradiation of adipocyte cells within the fat layer with sham BTL-9000 LLLT for the release of fat and lipids from these cells
  Arms: Placebo group

SUMMARY:
Prospective, two-arm, randomized study of the effectiveness of the BTL-9000 LLLT in achieving 3 cm or greater average waist circumferential reduction in LLLT group of subjects relative to the base line and 1 cm or greater reduction relative to the average waist circumferential reduction of the Placebo group.

DETAILED DESCRIPTION:
Prospective, randomized, blinded, two-arms study of waist circumferential reduction following 5 once-a-week treatments. One arm is the LLLT group of 25 subjects who are treated with the BTL-9000 LLLT and the other arm is the Placebo group of 15 subjects treated with the sham device. The objective of the study is to demonstrate the effectiveness of the BTL-9000 LLLT treatment in achieving average post-treatment waist circumferential reduction of 3 cm or greater across the waistline relative to the baseline assessment and of 1 cm or greater than the average waist circumferential reduction of the Placebo group.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18-70 years of age of both gender with excess adipose tissue in the abdomen area

  * Body Mass Index (BMI) of 25 to 35 kg/m2.
  * Subjects willing and able to abstain from partaking in any treatments other than the study procedure to promote body contouring and/or weight loss during study participation.
  * Subjects willing and able to maintain his/her regular (pre-procedure) diet and exercise regimen without effecting significant change in either direction during study participation.

Exclusion Criteria:

* Diabetics dependent on insulin or oral hypoglycemic medications
* Known cardiovascular disease such as arrhythmias, congestive heart failure
* Cardiac surgeries such as cardiac bypass, heart transplant surgery, pacemakers.
* Prior surgical interventions for body sculpting of abdomen such as liposuction
* Medical, physical or other contraindications for body sculpting/ weight loss
* Current use of medication known to affect weight levels and/or cause bloating or swelling and for which abstinence during the course of study participation is not safe or medically prudent
* Any medical condition known to affect weight levels and/or to cause bloating or swelling
* Active infection, wound or other external trauma to the area to be treated
* Pregnant, breast feeding, or planning pregnant before the end of the study
* Serious mental health illness
* Photosensitivity disorder to 660 nm light
* Active or recurrent cancer or current chemotherapy and/or radiation treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Waist Circumferential reduction | 30 days follow up after 8 twice-a-week treatments
  The subjects in the LLLT group whose average post-treatment waist circumference shows reduction of 3 cm or greater across the waistline relative to the base line assessment and their average waist circumferential reduction is 1 cm or greater than the average circumferential reduction of Placebo group are considered to meet the study primary outcome success criteria.

SECONDARY OUTCOMES:
Adverse Events | 1 month follow up
  Absence of adverse events (AE) associated with the treatment procedure. Safety evaluations of skin reaction in the treatment area would be conducted at every treatment and follow up visits

CONTACTS AND LOCATIONS:
Overall Officials: Radina Denkova, MD, Principal Investigator — Dermatologic Clinic